CLINICAL TRIAL: NCT03935646
Title: Acute Effects of Prescription Stimulant Medication on Cognition and Mood in College Students With and Without ADHD
Brief Title: Acute Effects of Stimulant Medication in College Students With ADHD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Cynthia M Hartung, PhD, Associate Professor, University of Wyoming
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190124JV02251
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Attention Deficit Hyperactivity Disorder; Stimulant Use; Working Memory; Change in Sustained Attention; Mood
Keywords: Attention Deficit Hyperactivity Disorder; Stimulant Use; Working Memory; Change in Sustained Attention; Mood
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This is a mixed (within-subjects and between-subjects) design. ADHD and comparison participants will complete outcome measures at baseline and at two counter-balanced experimental sessions (placebo, Adderall).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stimulant Medication (Experimental): Participants will be administered a stimulant medication (Adderall IR 10mg). The ordering of experimental vs. placebo appointments will be counterbalanced. Participants will complete computer-based tests of sustained attention and working memory during all appointments.
  Interventions: Drug: Adderall IR 10mg; Drug: Placebo

INTERVENTIONS:
Drug: Adderall IR 10mg — At one of the experimental appointments, participants will be administered a stimulant medication. Following a wait period, the participants will complete executive functioning tasks of working memory and sustained attention.
  Other Names: Stimulant Medication Manipulation
Drug: Placebo — Placebo

SUMMARY:
The investigators will examine the acute effects of stimulant medication on executive functioning. The rationale for the proposed study is to examine the efficacy of stimulants for college students with ADHD and help prevent stimulant misuse among college students without ADHD. The working hypothesis is that stimulants, compared to baseline and placebo conditions, will improve executive functioning for college students with ADHD but not for college students without ADHD. Improvements on executive functioning measures (e.g., CPT-IP, Spatial Span) will be examined through 2 (ADHD vs. non-ADHD) x 3 (Baseline, Placebo, Stimulant) repeated measures ANOVAs. Follow-up analyses will include paired comparisons.

Expected outcomes are to confirm these hypotheses and demonstrate the need for further study of stimulants. If confirmed, the results will provide pilot data for a larger NIH grant proposal aimed at further examining the acute effects of stimulants (i.e., improved cognitive functioning with stimulants) and comparing them to the acute effects of physical exercise (i.e., improved cognitive functioning immediately after exercise). The investigators expect this outcome to have an important positive impact because it can help support stimulant medication as an effective treatment for college students with ADHD (DuPaul et al., 2012). Additionally, demonstration that stimulants do not improve executive functioning for college students without ADHD can be used to help prevent and discourage stimulant misuse and diversion on college campuses (Hartung et al., 2013).

DETAILED DESCRIPTION:
Participants. The investigators will enroll 40 University of Wyoming (UW) and Laramie County Community College (LCCC) students including 20 with ADHD and 20 without ADHD (20 men, 20 women). Power analyses (G*Power 3.1; Faul et al., 2007) indicated a sample of at least this size is needed to provide 80% power to detect medium effects. Participants will be recruited through several means including targeted email announcements, flyers, and SONA pre-screener data.

Full exclusion criteria can be found in the "Eligibility" section below. Most notably, participants must stratify as being low risk for stimulant medication use. A health history screening questionnaire and additional health items will be used to screen participants and responses will be reviewed and approved by a medical consultant.

All prospective participants will attend a baseline appointment to confirm eligibility including: (a) being at low risk for stimulant use contraindications and (b) meeting diagnostic threshold for ADHD. After confirming eligibility, participants will also complete baseline measures during the baseline appointment. After enrolling in the study, participants will be scheduled for two experimental appointments. The two experimental appointments will include: (a) Placebo pill and (b) Stimulant (Adderall IR 10mg). The ordering of experimental appointments will be counterbalanced. Experimental appointments will be scheduled in the mornings and on the same day of the week and same time of day. Participants will be asked to abstain from caffeine, alcohol, nicotine, and illicit drugs for 12 hours prior to their appointments. Participants will be administered either placebo or stimulant. After a 90-minute wait, participants will complete executive functioning measures. Physiological measures (e.g., heart rate and blood pressure) will be monitored at specific times throughout the appointment and a medical consultant will be available on call for any emergencies. Participants will also be sent a modified mood (i.e., Depression, Anxiety, and Stress Scale or DASS) and sleep (Pittsburgh Sleep Quality Index or PSQI) questionnaire the morning following all experimental appointments. The only difference between the two appointments is the administration of either placebo or stimulant.

Prior to analyses, all variables will be screened. Violations of statistical assumptions will be addressed through data transformations or nonparametric statistics. Improvements on executive functioning measures (e.g., CPT-IP, Spatial Span) will be examined through 2 (ADHD vs. non-ADHD) x 3 (Baseline, Placebo, Stimulant) repeated measures ANOVAs. When interactions are significant, paired samples t-tests will be used to evaluate group differences. When interaction effects fail to reach statistical significance, independent samples t-tests will be used to evaluate group differences. The magnitude of omnibus effects for repeated measures ANOVAs will be calculated using partial eta-squared (ηp2). Within-group effects (Cohen's d) and corresponding confidence intervals for within-group effect sizes will be standardized using the variability of baseline scores (Howell, 2011). Between-group effects will be calculated using Hedges g (Hedges, 1982).

ELIGIBILITY:
Inclusion Criteria:

* Be currently enrolled either full time or part time as an undergraduate in a 2-year or 4-year college
* Be between the ages of 18-29
* Be a native English speaker
* ADHD Participants: Must report a prior diagnosis of ADHD and self-report five or more inattention (IA) symptoms on the DSM-5 Symptom Checklist on the pre-screener.
* Healthy Participants: Must disavow ever being diagnosed with ADHD, report 3 or fewer IA symptoms and 3 or fewer hyperactivity/impulsivity (HI) symptoms on the DSM-5 ADHD Symptom Checklist in the pre-screener and are an age and sex match of an ADHD group participant

Exclusion Criteria:

* Not meeting any of the above stated inclusion criteria
* Any contraindications for physical exercise placing the participant at moderate or high-risk. This includes the following:

  1. Participants will be excluded if they report having an acute or uncontrolled disease (cardiovascular, pulmonary, neurological, endocrine, musculoskeletal, immunological).
  2. Participants will be excluded if they are non-ambulatory or rely on walking aids for ambulation.
  3. Participants will be excluded who chronically manage asthma or another respiratory condition or require using an inhaler to complete exercise.
  4. Participants will be excluded if they experience uncontrolled or current problems with syncope (loss of consciousness or fainting) or postural hypotension.
  5. Participants will be excluded if they have ever had a stroke, aneurysm, or transient ischemic attack (TIA).
  6. Participants will be excluded if they have exercise or physical activity restrictions imposed by a health provider.
  7. Participants will be excluded by the medical director due to possible underlying disease/condition or risk.
  8. Participants will be excluded if they are pregnant (determined by a urine pregnancy test), are attempting to become pregnant, or are currently breastfeeding will also be excluded (stated above).
  9. Participants will be excluded for any current use of other psychotropic drugs (e.g., SSRIs, SNRIs, sedatives; stated above).
* Any contraindications for stimulant medication use placing the participant at moderate or high-risk. This includes the following:

  1. Participants will be excluded if they have ever been diagnosed with seizure disorder, high blood pressure, glaucoma, gastrointestinal hypermotility disorder (e.g., IBS), diabetes, hypoglycemia, cardiac problems (e.g., heart disease), or thyroid problems.
  2. Participants will be excluded if they have ever been diagnosed with a bipolar disorder (e.g., Bipolar I or Bipolar II), a psychotic disorder (e.g., schizophrenia), a sleep disorder (e.g., narcolepsy), an eating disorder (e.g., bulimia nervosa), or a severe substance use disorder (e.g., endorsing six or more symptoms of a substance use disorder according to the DSM-5). Participants will also be excluded if they report a past year diagnosis of major depressive disorder, panic disorder, generalized anxiety disorder, or any substance use disorder.
  3. Participants will be excluded if they report any prior treatment for substance use (e.g. rehabilitation for alcohol or other substance use). Additionally, participants will be excluded if they do not agree to abstain from illicit or addictive drugs and marijuana use for the duration of the study beginning with the eligibility assessment.
  4. Participants will be excluded if they experience uncontrolled or current problems with syncope (e.g., loss of consciousness or fainting) or postural hypotension.
  5. Participants will be excluded if they are pregnant (determined by a urine pregnancy test), are attempting to become pregnant, or are currently breastfeeding.
  6. Non-ADHD participants will be excluded if they have ever engaged in non-prescription stimulant use.
  7. ADHD participants who are currently prescribed a prescription stimulant will be asked not to take their medication the day prior to and day of any study visits. They will be excluded if they are not comfortable with abstaining.
  8. Participants will be excluded for any current use of other psychotropic drugs (e.g., SSRIs, SNRIs, sedatives) or non-stimulant ADHD medication (i.e., Strattera).
  9. Participants will be excluded for any current use of any other prescription medication that could interact negatively with Adderall (e.g., neurological and blood-pressure drugs, antihistamines).
  10. They will also be excluded for current use of high levels of caffeine consumption (e.g., daily use more than 600mg/day or about six 8-oz. cups of coffee). Daily use is defined as 5 or more days per week for the last month.
  11. Participants who are using other over-the-counter-substances that could interact negatively with Adderall (e.g., dietary supplements, weight-loss pills, and low-to-moderate levels of caffeine consumption, antihistamines) will be asked to abstain from use for at least 12-hours prior to lab visits. They will be excluded if they are not comfortable with abstaining.
  12. Participants will be excluded if they report current nicotine use (i.e., 5 or more cigarettes per day), daily vaping (i.e., e-cigarettes), smokeless tobacco (i.e., chewing tobacco), nicotine gum, and/or nicotine patches use in the past month.
  13. Participants will be excluded if they experienced a concussion within the past 6 months, have experienced two or more concussions in their lifetime, or have a history of traumatic brain injury.
  14. Participants will be excluded if they have ever had a stroke, aneurysm, or transient ischemic attack (TIA).
  15. Participants will be excluded if they are unwilling to ingest a prescription stimulant medication (Adderall) or placebo in the lab.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Continuous Performance Test - Identical Pairs (CPT-IP) for Adderall vs. Placebo | Completed at baseline and each experimental appointment over a period of three weeks
  The CPT-IP is a standardized computer-administered test consisting of four-digit numbers that are presented for 200ms on a white screen with 1500ms between the presentation of each number. Participants must press the spacebar as quickly as possible when the preceding four-digit number matches the current four-digit number. Participants will complete the CPT-IP as a measure of sustained attention at baseline and at each experimental appointment.
Change in Spatial Span (SS) for Adderall vs. Placebo | Completed at baseline and each experimental appointment over a period of three weeks
  The Spatial Span (SS) is a computer-administered task assessing visuospatial working memory. Participants will be tasked with remembering the order of stimuli that are presented in forward and backward sequences. Participants will complete the SS visuospatial working memory task at baseline and at each experimental appointment.
Change in Digit Span for Adderall vs. Placebo | Completed at baseline and each experimental appointment over a period of three weeks
  The Digit Span (Wechsler, 2008) subtest of the Wechsler Adult Intelligence Scale (WAIS-IV) is an auditory working memory task. The researcher will say numbers aloud at a rate of one number per second. The participant will be tasked with remembering and repeating the numbers in a prescribed (forward, backward, sequencing) order. Participants will complete the Digit Span (forward, backward and sequencing) auditory working memory task at baseline and at each experimental appointment.
Change in Letter-Number Sequencing for Adderall vs. Placebo | Completed at baseline and each experimental appointment over a period of three weeks
  The Letter-Number Sequencing (Wechsler, 2008) task is a supplemental subtest of the Wechsler Adult Intelligence Scale (WAIS-IV) that measures auditory working memory. Researchers will read a sequence of letters and numbers, and the participant will attempt to recall the numbers in ascending order and the letters in alphabetical order. Participants will complete the Letter-Number Sequencing auditory working memory task at baseline and at each experimental appointment.
Visual Analogue Scales (VAS) for Adderall vs. Placebo | two weeks
  The VAS is a nine-item questionnaire that assesses subjective mood in the moment including how good, bad, focused, and motivated participants feel. Additionally, participants are asked how well they expect to perform on cognitive tests and how much effort they will put into completing cognitive tests. Participants will complete the VAS at each experimental appointment.
Addiction Research Center Inventory (ARCI) for Adderall vs. Placebo | two weeks
  The ARCI is a 49 true-false item measure that assesses drug effects by asking how the participant feels in the moment. Participants will complete the ARCI at each experimental appointment.
Intentions to Use Questionnaire (IUQ) for Adderall vs. Placebo | two weeks
  The IUQ is a six-item measure that assesses the likelihood of participants to use substances including prescription stimulants for specific purposes such as for studying or improving academic performance. Participants will complete the IUQ at each experimental appointment.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index-Modified (PSQI-M) | Completed the day after each experimental appointment over a period of two weeks
  The PSQI contains 19 items that evaluates several components of sleep quality by requiring participants to report their sleep behaviors. Participants will receive the survey via text and email the morning after their experimental appointment. They will be instructed to complete the PSQI-M regarding their sleep functioning (i.e., subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction) from "yesterday (from the time after your lab appointment until you went to bed)."
Depression, Anxiety, and Stress Scale-Modified (DASS-M) | Completed the day after each experimental appointment over a period of two weeks
  This scale includes 21 questions to measure current mood and stress levels. Items include a choice of four responses from "Did not apply to me at all," to "Applied to me very much." Participants will receive the survey via text and email the morning after their experimental appointment. They will be instructed to complete the DASS-M regarding their emotional experiences of depression, anxiety, and stress from "yesterday (from the time after your lab appointment until you went to bed)."
DSM-5 ADHD Symptoms Checklist - Modified (DSM 5-M) | Completed the day after each experimental appointment over a period of two weeks
  The DSM 5-M will ask participants about how often they experienced the symptoms of ADHD for the 24 hours from "yesterday (from the time after your lab appointment until you went to bed)" and will be completed following both experimental sessions
Side Effects Rating Scale - Modified | Completed the day after each experimental appointment over a period of two weeks
  The Side Effects Rating Scale - Modified asks participants about behaviors from side effects of ADHD medication for the 24 hours from "yesterday (from the time after your lab appointment until you went to bed)" and will be completed following both experimental sessions
Substance Use Day After Questionnaire | Completed the day after each experimental appointment over a period of two weeks
  This Substance Use Day After Questionnaire asks participants if they engaged in any substance use (including use of alcohol, prescription stimulants, caffeine, cannabis, or other illicit substances) since "yesterday (from the time after your lab appointment until you went to bed)" and will be completed following both experimental sessions

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Hartung, Ph.D., Principal Investigator — University of Wyoming
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartung CM, Canu WH, Cleveland CS, Lefler EK, Mignogna MJ, Fedele DA, Correia CJ, Leffingwell TR, Clapp JD. Stimulant medication use in college students: comparison of appropriate users, misusers, and nonusers. Psychol Addict Behav. 2013 Sep;27(3):832-40. doi: 10.1037/a0033822. PMID 24059834
- [Background] Dupaul GJ, Weyandt LL, Rossi JS, Vilardo BA, O'Dell SM, Carson KM, Verdi G, Swentosky A. Double-blind, placebo-controlled, crossover study of the efficacy and safety of lisdexamfetamine dimesylate in college students with ADHD. J Atten Disord. 2012 Apr;16(3):202-20. doi: 10.1177/1087054711427299. Epub 2011 Dec 12. PMID 22166471